CLINICAL TRIAL: NCT01685099
Title: Evaluating the Diagnostic Validity of Inflammation-associated Markers for Tuberculous Pleurisy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207061RIC
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-08

CONDITIONS: To Investigate Diagnostic Aid of the Inflammation and Apoptosis-associated Markers and Apoptosis Pattern of PE Neutrophil for Tuberculous Pleurisy
Keywords: diagnosis, inflammation-associated markers, pleural effusion, tuberculosis, tuberculous pleurisy
MeSH Terms: conditions — Disease; Pleural Effusion; Tuberculosis; Tuberculosis, Pleural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pleural effusion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group with tuberculous pleurisy
- Group with non-tuberculous pleurisy

SUMMARY:
1. To investigate the difference of PE inflammation/apoptosis-associated markers between TB pleurisy and non-TB pleurisy
2. To investigate the difference of neutrophil apoptosis in exudative PE between TB pleurisy and non-TB pleurisy
3. To investigate the change of apoptosis pattern of PE neutrophil, before and after TB antigen stimulation, and compare the difference between TB pleurisy and non-TB pleurisy
4. To investigate diagnostic aid of the inflammation/apoptosis-associated markers and apoptosis pattern of PE neutrophil for tuberculous pleurisy

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a global health problem even though it has nearly been eradicated in some developed countries. Because of variable manifestations and the difficulty in collecting clinical samples, extra-pulmonary TB is usually difficult to early diagnose. Tuberculous pleurisy (TP) is one of the most common extra-pulmonary infection and accounts for approximately 5% of all forms of TB. The gold standard for diagnosing TP is mycobacterial culture of pleural effusion (PE), pleura tissue, which requires weeks to yield. The treatment could thus be delayed, resulting in an increased mortality rate. In addition, mycobacterial culture is not so sensitive for PE and with positivity in less than two thirds of cases with TB pleurisy.

For diagnosing TP, PE biomarkers are required to be investigated in addition to traditional PE cell counting and biochemistry. In particularly, inflammation-associated cytokines and apoptosis-associated markers may be important because the two pathways involve in TB infection/defense mechanism. For inflammation-association markers, current literature is not comprehensive except IFN-gamma and IFN-gamma release assay (IGRA). However, the result of IGRA using PE is disappointed. We should study other PE inflammation markers such as IFN-induced protein-10, interleukin [IL]-2, IL-12 and so on. On the other hand, apoptosis suppression is one of escape mechanisms in TB pathogenesis. Macrophage, dendritic cell, and neutrophil are reportedly inhibited for apoptosis in TB infection. But the apoptosis of PE neutrophil are rarely studied. Moreover, the role of apoptosis-associated markers (Fas ligand [FasL], decoy receptor 3, lipoxin, prostaglandin E2, caspases) in PE has rarely been investigated in diagnosing TP except FasL. Therefore, we conduct a prospective study to investigate inflammation/apoptosis-associated markers in exudative PE and apoptosis of PE neutrophil to analyze their diagnostic usefulness for TP.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 20 years old
* patients with exudative pleural effusion

Exclusion Criteria:

* refusal of enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with tuberculous pleural effusion
  2. Patients with pleural effusion due to causes other than tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08

PRIMARY OUTCOMES:
diagnosis of tuberculous pleurisy | 2 years

SECONDARY OUTCOMES:
mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan